CLINICAL TRIAL: NCT07072910
Title: Prevention and Treatment of Episodic Migraine by Cabergoline Therapy (PROTECT). A Randomized, Placebo-controlled, Double-blind, Investigator-initiated Trial
Brief Title: Cabergoline for Episodic Migraine
Acronym: PROTECT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AU-PROTECT-2025; 2025-522323-10-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-19; First posted 2025-07-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Migraine
Keywords: Migraine; Preventive treatment; Cabergoline; Drug repurposing
MeSH Terms: conditions — Migraine Disorders | interventions — Cabergoline; Dopamine Agonists

STUDY DESIGN:
Intervention Model Description: The PROTECT trial is a randomized, double-blind, placebo-controlled study. It includes:
  1. A baseline phase (Weeks -4-0): Participants complete a daily headache diary to document migraine frequency and classify headache days.
  2. A Double-Blind Phase (Weeks 0-12): Participants receive cabergoline 0.5 mg/week, cabergoline 1.0 mg/week, or placebo.
  3. An Open-Label Phase (Weeks 12-24): All participants receive cabergoline (0.5 mg or 1.0 mg) once weekly.
  4. A Safety Follow-Up Phase (Weeks 24-28): Participants are monitored for adverse events after discontinuation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cabergoline 0.5 mg/Week (Double-Blind Phase) (Experimental): Participants in this arm will receive cabergoline 0.5 mg once weekly as add-on treatment for 12 weeks during the double-blind treatment phase.
  Interventions: Drug: Cabergoline 0.5 MG
- Cabergoline 1.0 mg/Week (Double-Blind Phase) (Experimental): Participants in this arm will receive cabergoline 1.0 mg once weekly as add-on treatment for 12 weeks during the double-blind treatment phase.
  Interventions: Drug: Cabergoline 1 MG
- Placebo (Double-Blind Phase) (Placebo Comparator): Participants in this arm will receive a placebo once weekly as add-on treatment for 12 weeks during the double-blind treatment phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cabergoline 0.5 MG — Participants will receive cabergoline 0.5 mg as oral tablets, taken once weekly as an add-on treatment for 12 weeks during the double-blind treatment phase. Participants who received cabergoline 0.5 mg during the double-blind phase will continue with the same 0.5 mg dose in the open-label phase.
  Other Names: Dopamine receptor agonist; Dostinex
  Arms: Cabergoline 0.5 mg/Week (Double-Blind Phase)
Drug: Placebo — Participants will receive placebo as oral tablets, taken once weekly as an add-on treatment for 12 weeks during the double-blind treatment phase. In the open-label phase, these participants will transition to active cabergoline treatment, receiving either 0.5 mg or 1.0 mg once weekly, depending on their randomized allocation at the start of the open-label phase. The placebo tablets will be formulated to match the cabergoline tablets in size, shape, and color, and should be taken under the same conditions.
  Arms: Placebo (Double-Blind Phase)
Drug: Cabergoline 1 MG — Participants will receive cabergoline 1.0 mg as oral tablets, taken once weekly as an add-on treatment for 12 weeks during the double-blind treatment phase. Participants who received cabergoline 1.0 mg during the double-blind phase will continue with the same 1.0 mg dose in the open-label phase.
  Other Names: Dopamine receptor agonist; Dostinex
  Arms: Cabergoline 1.0 mg/Week (Double-Blind Phase)

SUMMARY:
The goal of this randomized, placebo-controlled, double-blind clinical trial is to evaluate the efficacy, safety, and tolerability of cabergoline for the prevention of episodic migraine in adults with 4-14 monthly migraine days (MMD). The main questions it aims to answer are:

1. Does once-weekly cabergoline (0.5 mg or 1.0 mg) reduce MMD compared to placebo?
2. What are the effects of cabergoline on headache severity, acute medication use, and patient-reported outcomes?
3. Is cabergoline safe to use in individuals with migraine?

Participants will:

Complete a 4-week baseline period to document migraine frequency and classify headache days.

Be randomly assigned to one of three treatment arms:

1. Cabergoline 0.5 mg/week
2. Cabergoline 1.0 mg/week
3. Placebo

Participate in a 12-week double-blind treatment phase, followed by a 12-week open-label treatment phase where all participants receive cabergoline (0.5 mg or 1.0 mg once weekly).

Record daily headache activity, acute medication use, and severity using an electronic diary.

Complete validated headache questionnaires and provide blood samples for biomarker analysis at baseline, week 12, and week 24.

The study also includes exploratory analyses of genetic predictors of treatment response and metabolic markers to assess the broader effects of cabergoline.

DETAILED DESCRIPTION:
Migraine is a common and often disabling neurological disorder. While there are several treatments available, many individuals continue to experience frequent attacks, side effects from medications, or limited access to newer therapies due to high costs.

Cabergoline is a medication that activates dopamine receptors and has shown promising effects in migraine. A small, pilot study found that a low dose of cabergoline (0.5 mg per week) reduced the number of migraine days per month in patients with episodic migraine. It was well tolerated, with few side effects and good treatment adherence.

The PROTECT trial is a larger clinical study that aims to confirm these results. The trial will evaluate whether cabergoline, taken once weekly, is effective in reducing the number of monthly migraine days compared to placebo. It will also test a higher dose (1.0 mg/week) to investigate whether a stronger effect can be achieved without increasing side effects.

The trial consists of two treatment phases. In the first phase, participants will be randomly assigned to receive either cabergoline 0.5 mg, cabergoline 1.0 mg, or placebo once weekly for 12 weeks. In the second phase, all participants will receive cabergoline for another 12 weeks, in an open-label setting. This will allow researchers to study longer-term treatment effects, adherence, and tolerability. A final safety follow-up phase will last four weeks.

Throughout the study, participants will report their migraine symptoms, medication use, and headache severity in a secure electronic diary. They will also complete questionnaires about headache-related disability, work productivity, and overall improvement. Blood samples will be collected to study the underlying biological mechanisms of migraine, and explore whether certain genetic or hormonal markers can help predict who benefits most from cabergoline.

The main outcome of the study is the change in the number of monthly migraine days during the last four weeks of the double-blind phase. Other outcomes include changes in headache severity, use of acute medication, and quality-of-life scores. The study will also monitor changes in health markers such as cholesterol, inflammation, and prolactin levels.

The PROTECT trial will include adults with episodic migraine (defined as having 4 to 14 migraine days per month). Participants must be at least 18 years old and have had a stable pattern of migraine attacks and acute treatment for the past three months. People with chronic migraine, certain headache types, or other medical conditions will not be eligible.

Participants will be recruited from headache clinics, general practitioners, and online platforms. All participants will provide written informed consent before entering the study.

This trial is conducted by an independent academic research group and is designed to evaluate a low-cost, well-known medication for a new use. If successful, cabergoline could provide a new, accessible preventive option for people with migraine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Episodic migraine according to ICHD-3 criteria
* 4-14 monthly migraine days (MMD) in the last 3 months prior to inclusion
* Stable acute migraine medication use for at least 3 months prior to inclusion
* Written informed consent

Exclusion Criteria:

* < 4 MMD or ≥ 15 MMD during the baseline period
* Chronic migraine (≥15 headache days per month)
* Trigeminal autonomic cephalalgias and neuralgias
* Secondary headache conditions
* Other common primary headache types (e.g. tension-type headache) if attacks are frequent (present on an average of >1 day/month and >12 days/year)
* Presumed medication-overuse headache
* Recent changes in preventive migraine treatment (≥3 months prior to study inclusion)
* History of pulmonary, retroperitoneal, or pericardial disorders, including heart valve disease
* Severe untreated hypertension
* Use of drugs with dopamine antagonistic or agonistic properties
* Psychiatric disorders requiring pharmacological treatment
* Women of child-bearing potential (i.e. not chemically or surgically sterilized, or not postmeno-pausal) and male participants with partners of child-bearing potential, who are unwilling to use a medically accepted method of contraception, considered reliable by the investigator, from signing of informed consent and throughout the study
* Women who have a positive pregnancy test at randomization
* Women who are breast-feeding
* Allergy or hypersensitivity to cabergoline or similar compounds
* Concurrent participation in another clinical trial that, in the judgement of the investigator, may interfere with the conduct or outcomes of the present study
* Inability of the subject, in the opinion of the investigator, to understand and/or comply with study medications or procedures, or any conditions that, in the opinion of the investigator, may render the subject unable to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Monthly Migraine Days (MMD) | Baseline to the last four weeks of the double-blind treatment phase
  Change in MMD from baseline to the last four weeks of the double-blind treatment phase.
  Migraine days are defined according to ICHD-3 criteria or the use of migraine-specific acute medication, recorded in a daily, electronic diary.

SECONDARY OUTCOMES:
Responder rate (proportion of participants achieving ≥50% reduction in MMD) | Baseline to the last four weeks of the double-blind treatment phase.
  Proportion of participants achieving ≥50% reduction in MMD during the last four weeks of the 12-week double-blind treatment phase (50% responder rate).
Change in number of moderate/severe headache days | Baseline to the last four weeks of the double-blind treatment phase.
  Change in number of moderate/severe headache days from baseline to the last four weeks of the double-blind treatment phase.
Headache severity | The last four weeks of the double-blind treatment phase.
  Proportion of attacks classified as mild, moderate, or severe at the last four weeks of the double-blind treatment phase.
Changes in acute medication use. | Baseline to the last four weeks of the double-blind treatment phase.
  Change in number of days with use of acute migraine-specific medication from baseline to the last four weeks of the double-blind treatment phase.
Migraine Disability Assessment Scale (MIDAS) | Baseline to the end of the double-blind treatment phase (week 12).
  Change in MIDAS score from baseline to the end of the double-blind treatment phase. MIDAS assesses migraine-related disability over a 3-month recall period. It contains five questions regarding number of days of missed work/school, reduced productivity at work/school, missed household work, reduced productivity in household work, and missed family and/or social activities. A higher score indicates greater disability.
Headache Impact Test - 6 items (HIT-6) | Baseline to the end of the double-blind treatment phase (week 12).
  Change in HIT-6 score from baseline to the end of the double-blind treatment phase. HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. A higher score indicates greater disability.
Work Productivity and Activity Impairment (WPAI) | Baseline to the end of the double-blind treatment phase (week 12).
  Change in WPAI score from baseline to the end of the double-blind treatment phase. WPAI Questionnaire is a 6-item instrument to measure impairments over the past 7 days in both paid work and unpaid work due to one's health. A higher score indicates greater disability.
Patient's Global Impression of Change (PGIC) | The end of the double-blind treatment phase (Week 12)
  PGIC score at the end of the double-blind treatment phase.
Safety and tolerability of cabergoline (incidence of adverse events) | From the beginning of the treatment phase (week 0) until the end of the safety follow-up (week 28).
  Incidence of adverse events during the trial.
Sustained effect of cabergoline treatment in change in MMD. | Baseline to the last four weeks of the open-label phase, and from the last four weeks of the double-blind phase to the last four weeks of the open-label phase.
  Change in MMD assessed from baseline and from the end of the double-blind phase to the end of the open-label phase.
Sustained effect of cabergoline on responder rate (defined as the proportion of participants achieving a ≥50% reduction in monthly migraine days). | Baseline to the last four weeks of the open-label phase, and from the last four weeks of the double-blind phase to the last four weeks of the open-label phase.
  Proportion of participants achieving ≥50% reduction in MMD assessed from baseline and from the end of the double-blind phase to the end of the open-label phase.
Sustained effects of cabergoline on the frequency of moderate/severe headache days. | Baseline to the last four weeks of the open-label phase, and from the last four weeks of the double-blind phase to the last four weeks of the open-label phase.
  Number of moderate/severe headache days assessed from baseline and from the end of the double-blind phase to the end of the open-label phase.
Sustained effects of cabergoline treatment on acute medication use. | Baseline to the last four weeks of the open-label phase, and the last four weeks of the double-blind phase to the last four weeks of the open-label phase.
  Acute medication use assessed from baseline and from the end of the double-blind phase to the end of the open-label phase.
Sustained effects of cabergoline treatment on HIT-6 score. | Baseline to the last four weeks of the open-label phase, and the last four weeks of the double-blind phase to the last four weeks of the open-label phase.
  Change in HIT-6 score from baseline and from the end of the double-blind phase to the end of the open-label phase.
Sustained effects of cabergoline treatment on MIDAS score. | Baseline to the last four weeks of the open-label phase, and the last four weeks of the double-blind phase to the last four weeks of the open-label phase.
  Change in MIDAS score from baseline and from the end of the double-blind phase to the end of the open-label phase.
Sustained effects of cabergoline treatment on WPAI score. | Baseline to the last four weeks of the open-label phase, and the last four weeks of the double-blind phase to the last four weeks of the open-label phase.
  Change in WPAI score from baseline and from the end of the double-blind phase to the end of the open-label phase.
Sustained effects of cabergoline treatment on PGIC. | The end of the double-blind phase (week 12) and the end of the open-label phase (week 24).
  PGIC (participant's overall perception of change since starting study medication) assessed at the end of the double-blind phase compared to the end of the open-label phase.
Comparison of any treatment (0.5 mg or 1.0 mg) versus placebo on MMD | Baseline to the last four weeks of the double-blind treatment phase.
  Change in MMD from baseline to the last four weeks of the double-blind phase in any treatment (0.5 mg or 1.0 mg) versus placebo.
Comparison of any treatment (0.5 mg or 1.0 mg) versus placebo on responder rate | Baseline to the last four weeks of the double-blind treatment phase.
  Proportion of participants achieving ≥50% reduction in MMD in the group receiving cabergoline (0.5 mg or 1.0 mg) compared to placebo from baseline to the last four weeks of the double-blind phase.
Comparison of any treatment (0.5 mg or 1.0 mg) versus placebo on number of moderate/severe headache days | Baseline to the last four weeks of the double-blind treatment phase.
  Number of moderate/severe headache days with any treatment (0.5 mg or 1.0 mg) versus placebo from baseline to the last four weeks of the double-blind phase.
Comparison of any treatment (0.5 mg or 1.0 mg) versus placebo on acute medication use | Baseline to the last four weeks of the double-blind treatment phase.
  Acute medication use with any treatment (0.5 mg or 1.0 mg) versus placebo from baseline to the last four weeks of the double-blind phase.
Comparison of any treatment (0.5 mg or 1.0 mg) versus placebo on HIT-6 | Baseline to the last four weeks of the double-blind treatment phase.
  HIT-6 score with any treatment (0.5 mg or 1.0 mg) versus placebo from baseline to the last four weeks of the double-blind phase.
Comparison of any treatment (0.5 mg or 1.0 mg) versus placebo on MIDAS | Baseline to the last four weeks of the double-blind treatment phase.
  MIDAS score with any treatment (0.5 mg or 1.0 mg) versus placebo from baseline to the last four weeks of the double-blind phase.
Comparison of any treatment (0.5 mg or 1.0 mg) versus placebo on WPAI | Baseline to the last four weeks of the double-blind treatment phase.
  WPAI with any treatment (0.5 mg or 1.0 mg) versus placebo from baseline to the last four weeks of the double-blind phase.
Comparison of any treatment (0.5 mg or 1.0 mg) versus placebo on PGIC | The end of the double-blind treatment phase (week 12).
  PGIC (participant's overall perception of change since starting study medication) with any treatment (0.5 mg or 1.0 mg) versus placebo after the double-blind treatment phase.
Dose-Response Analysis of Change in Monthly Migraine Days (MMD) | Baseline to the last four weeks of the double-blind treatment phase.
  Monthly Migraine Days (MMD) will be assessed as the change from baseline to the last four weeks of the double-blind phase. MMD is defined as the number of migraine days per 28-day period, recorded via electronic headache diary. The dose-response relationship will be evaluated by comparing the change in MMD across the three treatment arms (placebo, cabergoline 0.5 mg, and cabergoline 1.0 mg) in a single model.
Dose-Response Analysis of ≥50% Responder Rate in Monthly Migraine Days. | Baseline to the last four weeks of the double-blind treatment phase.
  Responder rate is defined as the proportion of participants achieving a ≥50% reduction in Monthly Migraine Days (MMD) from baseline to the last four weeks of the double-blind phase. MMD is measured as the number of migraine days per 28-day period, recorded via electronic headache diary. The dose-response relationship will be assessed by comparing responder rates across the three treatment arms (placebo, cabergoline 0.5 mg, and cabergoline 1.0 mg) in a single model.
Dose-Response Analysis of Moderate/Severe Headache Days | Baseline to the last four weeks of the double-blind treatment phase.
  Moderate/severe headache days will be assessed as the number of days per 28-day period with a headache rated as moderate or severe in intensity, based on daily entries in an electronic headache diary. A dose-response relationship will be evaluated by comparing moderate/severe headache days across the three treatment arms (placebo, cabergoline 0.5 mg, and cabergoline 1.0 mg) in a single model. The outcome is defined as the change from baseline to the last four weeks of the double-blind phase.
Dose-Response Analysis of Acute Migraine Medication Use | Baseline to the last four weeks of the double-blind treatment phase.
  Acute medication use is defined as the number of days per 28-day period on which any acute migraine-specific medication (e.g., triptans or gepants) is used, based on entries in an electronic headache diary. The outcome is assessed as the change from baseline to the last four weeks of the double-blind phase. A dose-response relationship will be evaluated by comparing acute medication use across the three treatment arms (placebo, cabergoline 0.5 mg, and cabergoline 1.0 mg) in a single model.
Dose-Response Analysis of HIT-6 Total Score | Baseline to the last four weeks of the double-blind treatment phase.
  The Headache Impact Test-6 (HIT-6) assesses the impact of headache on daily functioning, including pain, social functioning, and cognitive performance. The total score ranges from 36 to 78, with higher scores indicating greater headache-related disability. The outcome is defined as the change in HIT-6 total score from baseline to the last four weeks of the double-blind phase. A dose-response relationship will be evaluated by comparing HIT-6 score changes across the three treatment arms (placebo, cabergoline 0.5 mg, and cabergoline 1.0 mg) in a single model.
Dose-Response Analysis of MIDAS Total Score | Baseline to the last four weeks of the double-blind treatment phase.
  The Migraine Disability Assessment (MIDAS) questionnaire evaluates headache-related disability over a 3-month period. Higher scores indicate greater disability. The outcome is defined as the change in MIDAS total score from baseline to the last four weeks of the double-blind phase. A dose-response relationship will be evaluated by comparing changes in MIDAS score across the three treatment arms (placebo, cabergoline 0.5 mg, and cabergoline 1.0 mg) in a single model.
Dose-Response Analysis of Total WPAI (Migraine) Score | Baseline to the last four weeks of the double-blind treatment phase.
  The Work Productivity and Activity Impairment Questionnaire - Migraine version (WPAI:Migraine V2.0) is a validated instrument assessing the impact of migraine on work productivity and daily activities over the past seven days. The total score combines absenteeism, presenteeism, and activity impairment into a composite percentage ranging from 0% (no impairment) to 100% (complete impairment). The outcome is defined as the change in total WPAI score from baseline to the last four weeks of the double-blind phase. A dose-response relationship will be evaluated by comparing total scores across the three treatment arms (placebo, cabergoline 0.5 mg, and cabergoline 1.0 mg) in a single model.
Dose-Response Analysis of Patient Global Impression of Change (PGIC) | Baseline to the last four weeks of the double-blind treatment phase.
  The Patient Global Impression of Change (PGIC) is a single-item patient-reported outcome measuring the participant's overall perception of change in their condition since the start of study treatment. The outcome is defined as the PGIC score at the end of the double-blind phase. A dose-response relationship will be evaluated by comparing PGIC scores across the three treatment arms (placebo, cabergoline 0.5 mg, and cabergoline 1.0 mg) in a single model.

OTHER OUTCOMES:
Pharmacogenetic predictors of treatment response. | Baseline
  Genotyping of all participants for variants in the prolactin receptor and dopaminergic pathways previously associated with migraine and drug response.
Cost-effectiveness. | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Estimation of cost per responder and cost per QALY gained. This analysis will be descriptive and exploratory.
Change in serum prolactin. | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Change in serum prolactin levels from baseline to the end of the double-blind and open-label treatment phases. Descriptive analyses will be performed, and potential associations between prolactin levels and treatment response will be explored.
Exploratory Subgroup Analyses of Efficacy Outcomes | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Stratified analyses of pre-specified efficacy outcomes (e.g., MMD, responder rate, acute medication use, HIT-6, MIDAS, WPAI, PGIC) will be conducted by subgroups including sex, menopausal status, migraine with/without aura, presence of dopaminergic symptoms, and number of prior preventive treatments. These analyses are exploratory and intended to assess consistency of treatment effects across clinically relevant subgroups.
Incidence of adverse events (AEs) in relevant subgroups. | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Stratified analyses of incidence of AEs by sex, menopausal status, aura, presence of dopaminergic symptoms, and number of prior preventive treatments.
LDL | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Change in LDL from baseline to the end of the double-blind and open-label phases.
hs-CRP | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Change in hs-CRP from baseline to the end of the double-blind and open-label phases.
HbA1c | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Change in HbA1C from baseline to the end of the double-blind and open-label phases.
HDL | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Change in HDL from baseline to the end of the double-blind and open-label phases.
Total cholesterol | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Change in total cholesterol from baseline to the end of the double-blind and open-label phases.
Triglycerides | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Change in triglycerides from baseline to the end of the double-blind and open-label phases.
FSH | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Change in FSH from baseline to the end of the double-blind and open-label phases.
LH | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Change in LH from baseline to the end of the double-blind and open-label phases.
Estrogen/testosterone | Baseline to the end of the double-blind phase (week 12) and the end of the the open-label phase (week 24).
  Change in estrogen/testosterone from baseline to the end of the double-blind and open-label phases.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with researchers upon reasonable request, including baseline characteristics, outcome measures, and adverse events. Data will be available upon publication of the primary manuscript and for a minimum of 5 years. Requests should be directed to the Principal Investigator at ajh@clin.au.dk. Access will be granted upon approval of a data sharing agreement
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified individual participant data (IPD) and supporting information will be available upon publication of the primary manuscript and for a minimum of 5 years thereafter.
Access Criteria: Access to IPD and supporting documents will be granted to qualified researchers upon reasonable request, subject to approval of a data sharing agreement. Requests should be directed to the Principal Investigator at ajh@clin.au.dk. Researchers must provide a sound scientific proposal and agree to use the data only for the purpose described in the approved data sharing agreement.

REFERENCES:
- [Background] Hjelholt AJ, Bach FW, Kasch H, Stovring H, Jensen TS, Jorgensen JOL. Cabergoline as a preventive migraine treatment: A randomized clinical pilot trial. PLoS One. 2025 Apr 1;20(4):e0320937. doi: 10.1371/journal.pone.0320937. eCollection 2025. PMID 40168298